CLINICAL TRIAL: NCT04190121
Title: Perioperative Nutritional Support in Esophageal Cancer Patients
Acronym: NEEC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: THEODOROU DIMITRIOS (Other)
Responsible Party: Sponsor-Investigator, THEODOROU DIMITRIOS, PROFESSOR, University of Athens
Organization: University of Athens (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17771
Record Dates: First submitted 2019-12-04; First posted 2019-12-09 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Esophageal Cancer; Nutritional Deficiency
Keywords: esophageal cancer,nutritional support
MeSH Terms: conditions — Esophageal Neoplasms; Malnutrition

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP A (Experimental)
  Interventions: Dietary Supplement: prosure
- GROUP B (No Intervention)

INTERVENTIONS:
Dietary Supplement: prosure — The study group will receive the dietary supplement preoperatively and for three months after the operation
  Arms: GROUP A

SUMMARY:
Upper GI malignancies often lead to involuntary weight loss and nutritional deficits. Nutritional support, both pre- and postoperatively, may improve post-operative course and reduce length of hospital stay. This prospective randomized trial aims to investigate the above mentioned hypothesis and clarify any variants that may differ between the investigation and control group at a statistically significant level.

DETAILED DESCRIPTION:
This prospective randomized trial is conducted in the 1st Propaedeutic Department of Surgery of National and Kapodistrian University of Athens. The study population consists of adults suffering from upper GI malignancy. Informed consent is obtained in written. Following this, the patient is classified in either the intervention group or the control group. Patients belonging in the control group will receive the usual postoperative care, while the patients in the intervention group will receive nutritional support perioperatively. The aforementioned "usual postoperative care" consists of administration of intravenous fluids until resuming oral feeding, jejunostomy feeding starting from the first postoperative day, epidural analgesics for the first four postoperative days, perioperative administration of a second generation cephalosporin plus metronidazole and thromboprophylaxis with (low moleculr weight heparin (LMWH). The patients are also receiving appropriate for any concomitant health problems (e.g. existing diabetes mellitus) and transfusions based on their needs. We record the patient's age, the stage and histologic type of the disease, administration of adjuvant and/or neoadjuvant therapy and the patient's American Society of Anesthesiologists Score. Their preoperative nutritional state will be assessed using Body Mass Index (BMI), serum albumin, body fat percentage, muscle mass and total body water following measurement with body composition analyzer (Tanita MC-780U Multi Frequency Segmental Body Composition Analyzer). At their initial assessment the patients will fill in an appropriate quality of life questionnaire. The type of the operation, the use of drains and catheters, the patients needs in iv fluids, blood product transfusions, sedatives and analgesics during the operation will also be recorded. The postoperative course of any patient will be closely monitored, including the postoperative needs in fluid administration and analgesics, the need for transfusion, the administration of perioperative antibiotics, the removal of drains and catheters, the time of first bowel movement,the need of ICU hospitalization, the total length of hospital stay as well as any in-hospital complications. Upon discharge from the hospital, the control group will receive instructions on oral and jejunostomy feeding, while the intervention group will receive additional nutritional support for 3 months. Both patient groups will undergo post-operative follow-up for six months. In the first, third and sixth postoperative month body weight and its change, BMI, serum albumin, body fat percentage, muscle mass and total body water, as well as quality of life, postoperative complications and need for readmission will be evaluated. Neoadjuvant therapy will also be taken into account. The results will be statistically evaluated after appropriate stratification.

ELIGIBILITY:
Inclusion Criteria:

* patients with esophageal cancer
* 18 years or older

Exclusion Criteria:

-none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2019-03-26 (Actual); Primary Completion 2022-02-14 (Estimated); Study Completion 2022-02-14 (Estimated)

PRIMARY OUTCOMES:
infective complications | first six postoperative months
  surgical site infection,pneumonia,intraabdominal sepsis,postoperative fever or other signs of sepsis

SECONDARY OUTCOMES:
anastomotic leak | first six postoperative months
  anastomotic leak confirmed either by a CT scan or upper gastrointestinal series
postoperative arrhythmia or other cardiac complications | first six postoperative months
  cardiac complications confirmed by ECG that required consultation by a cardiologist
readmission rate | first six postoperative months
reoperation | first six postoperative months
  need for reoperation due to postoperative complications in the first six postoperative months
disease-associated death during the first six postoperative months | first six postoperative months
  death related to the known malignancy,including postoperative complications
length of hospital stay | first six postoperative months (including first admission and any other readmission)
  postoperative duration of hospital stay
length of stay in the ICU | first six postoperative months

OTHER OUTCOMES:
patient's BMI changes | first six postoperative months
patient's muscle mass changes | first six postoperative months
patient's body fat changes | first six postoperative months
patient's serum albumin changes | first six postoperative months

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Theodorou, Study Chair — Hippocration Hospital; Athina-Despina Kimpizi, Principal Investigator — Hippocration Hospital
Locations (1):
- Hippocration Hospital, Athens, Greece